CLINICAL TRIAL: NCT01635348
Title: Benefits of Two Types of Therapeutic Exercise on Gait and Cognition
Brief Title: Thinking, Walking Outcomes by Type of Exercise
Acronym: 2-STEP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO10090070; P30AG024827 (NIH)
Record Dates: First submitted 2012-06-22; First posted 2012-07-09 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2012-06

CONDITIONS: Gait Disorder, Sensorimotor; Cognitive Disorder
Keywords: gait speed; cognitive processing speed
MeSH Terms: conditions — Gait Disorders, Neurologic; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- motor skill gait exercise arm (Experimental): motor skill gait exercise intervention: stepping and walking patterns, and speed interval treadmill-assisted walking to enhance timing and coordination in walking
  Interventions: Behavioral: motor skill gait exercise
- aerobic gait exercise arm (Active Comparator): aerobic gait exercise intervention: treadmill-assisted and overground walking exercise to enhance walking practice and improve endurance in walking
  Interventions: Behavioral: aerobic gait intervention

INTERVENTIONS:
Behavioral: motor skill gait exercise — The motor skill gait exercise is a task-oriented motor sequence learning approach to exercise to improve walking. The approach involves goal-directed stepping and walking patterns to facilitate use of the appropriate muscles at the appropriate timing relative to body position during gait through the task performance. Treadmill-assisted walking in brief intervals of small increased speed walking interspersed with usual walking speed are performed to induce the automatic rhythm and timing of gait. The exercise sessions are about 60 minutes, 2-3 times a week for 12 weeks or a total of 30-36 sessions.
  Other Names: task-oriented motor sequence gait exercise; motor learning gait exercise; timing and coordination therapeutic gait activity
  Arms: motor skill gait exercise arm
Behavioral: aerobic gait intervention — The aerobic gait intervention approach involves treadmill and overground walking with the gradual increases in the distance walked and speed of walking. The exercise approach provides walking practice, including on the treadmill to facilitate the timing of stepping during gait, while also facilitating a fitness or conditioning response, and endurance for walking activities. The exercise sessions are about 60 minutes, 2-3 times weekly for 12 weeks, or about 30-36 sessions.
  Other Names: walking endurance exercise; aerobic walking training; impairment-oriented gait exercise
  Arms: aerobic gait exercise arm

SUMMARY:
The purpose of this research study is to compare two different exercise treatments for walking problems in older adults. The investigators want to determine if participation in the exercise programs will improve walking and thinking abilities.

DETAILED DESCRIPTION:
Specific Aims We will examine the impact of moderate intensity aerobic and of motor skill exercise interventions on improving gait and cognition in older adults with slow gait and psychomotor slowing. In a thrice weekly, 12 week, randomized clinical trial, we propose the following aims: 1) to define the impact of moderate intensity aerobic and motor skill gait exercise on thinking while walking, and 2) to define the impact of moderate intensity aerobic and motor skill gait exercise on gait and cognition. Brief Background The optimal exercise to improve gait and brain health in older adults is not known. Two types of exercise with potential for affects on gait and brain health, aerobic and motor skill exercise, developed out of distinct disciplines and have been studied separately, but not in older adults with the same age-related, centrally-generated slow gait dysfunction or for their effects on an integrated measure of gait and cognition, 'walking while thinking'. Summary of Methods We propose two parallel, single arm clinical trials to define the impact of aerobic and motor-skill exercise on gait and cognitive functions, in community-dwelling older adults with slow gait and psychomotor slowing, randomly assigned to moderate intensity aerobic gait (n=12) or motor skill gait (n=12) exercise, three times a week, for 12 weeks, in small groups of 2-3 supervised by a physical therapist. Primary outcomes are integrated measures of thinking while walking, with secondary outcomes of specific measures of gait and cognitive function collected pre, 4, 8 and 12 weeks post interventions, to examine impact of exercise and dose-response effects on gait and cognition. Future Use of Data The intent of the proposed pilot is to generate complementary data essential to support an R01 clinical trial grant submission. Specifically in this pilot we will: 1) recruit older adults with both slow gait speed and evidence of psychomotor slowing, 2) explore and define a primary outcome measure that integrates both gait and cognition, and thus better represents the goal of the exercise interventions - thinking while walking, 3) determine potential mean and variability estimates for gait and cognitive outcomes, particularly the less well-characterized gait outcomes of aerobic exercise (energy expenditure for walking, gait variability, gait abnormalities), and cognitive outcomes of motor skill exercise (speed of processing, executive function).

ELIGIBILITY:
Inclusion Criteria:

* slow gait speed (<= 1.0m/s and >= .6m/s)
* slow cognitive processing (digit symbol substitution < age-adjusted norm
* medical clearance from primary physician for participation in exercise

Exclusion Criteria:

* dementia or Mild Cognitive Impairment MCI
* pain while walking that limits walking
* active medical conditions, not controlled or managed

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-01; Primary Completion 2013-05 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
integrated measure of thinking while walking | 12 weeks
  The outcome measure is a cognitive task such as working memory, visual-spatial orientation, and set shifting measures of cognitive function performed while walking over an oval track.

SECONDARY OUTCOMES:
gait | 12 weeks
  energy cost of walking, gait smoothness, gait speed and spatial and temporal gait characteristics under usual and challenging gait conditions, gait abnormalities, and walking endurance

CONTACTS AND LOCATIONS:
Overall Officials: Jessie M VanSwearingen, PhD, PT, Principal Investigator — University of Pittsburgh, Department of Physical Therapy
Locations (1):
- University of Pittsburgh, Department of Physical Therapy, Pittsburgh, Pennsylvania, United States